CLINICAL TRIAL: NCT01908218
Title: The Reliability and Validity of the Upper Lip Bite Test to Predict Difficult Laryngoscopy in Korean
Status: Completed | Type: Observational
Sponsor: Yonsei University (Other)
Responsible Party: Sponsor
Other Study IDs: 4-2008-0583
Record Dates: First submitted 2013-07-17; First posted 2013-07-25 (Estimated); Last update posted 2013-07-25 (Estimated); Status verified 2013-07

CONDITIONS: Orotracheal Intubation
Keywords: ULBT, diffficult laryngoscopy, Predictive Value of Tests

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- ULBT group: 344 adult patients undergoing general anesthesia with orotracheal intubation

SUMMARY:
Anticipated difficulties at laryngoscopy give time to prepare alternative method and proper management.

Several methods to evaluate the anatomical structures has been used during preoperative period for airway assessment.

Evaluation methods are such as the Mallampati classification, mouth opening, thyromental distance and sternocostal distance.

the Upper Lip Bite test, evaluates the possibility of a patient cover the mucosa of the upper lip by the lower incisor.

The aim of this study was to assess the clinical usefulness of the Upper Lip Bite test(ULBT) in Korean compared to Modified Mallampati classification(MMT).

ELIGIBILITY:
Inclusion Criteria:

* adult patients undergoing general anesthesia with orotracheal intubation

Exclusion Criteria:

* patient who have facial anomaly , 2. patients who required a rapid sequence induction

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: adult patients undergoing general anesthesia with orotracheal intubation
Sampling Method: Non-Probability Sample
Enrollment: 344 (Actual)
Dates: Start 2009-02; Primary Completion 2009-02 (Actual); Study Completion 2009-02 (Actual)

PRIMARY OUTCOMES:
Cormack and Lehane grade | glottis view with direct laryngoscopy for 1 minute during anesthesia induction
  When the patients undergoing general anesthesia with orotracheal intubation, after obtained glottis view with direct laryngoscopy, the performer assessed Cormack and Lehane grade. (It takes about 1 minutes). A grade 1 and 2 were rated as an easy laryngoscopy. Difficult laryngoscopy was defined as the inability to visualize the vocal cords, each includes Grades 3 and 4.

CONTACTS AND LOCATIONS:
Locations (1):
- Kwandong university colloge of medicine, Seoul, Seoul, South Korea

REFERENCES:
- [Derived] Kim JC, Ki Y, Kim J, Ahn SW. Ethnic considerations in the upper lip bite test: the reliability and validity of the upper lip bite test in predicting difficult laryngoscopy in Koreans. BMC Anesthesiol. 2019 Jan 10;19(1):9. doi: 10.1186/s12871-018-0675-5. PMID 30630419